CLINICAL TRIAL: NCT07186452
Title: A Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of HS-20093 in Patients With Advanced Solid Tumors Who Have Failed Adequate Standard Treatments or Are Intolerant to Standard Therapies
Brief Title: Evaluation of the Effect of Itraconazole on the Pharmacokinetics of HS-20093 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-111
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HS-20093 + Itraconazole (Experimental)
  Interventions: Drug: HS-20093; Drug: Itraconazole

INTERVENTIONS:
Drug: HS-20093 — All participants will receive intravenous infusion of HS-20093 at a dose of 8 mg/kg every 3 weeks (Q3W), with each treatment cycle lasting 21 days.
Drug: Itraconazole — Participants will then take itraconazole capsules orally at 200 mg per dose during C2D17-C3D21

SUMMARY:
The primary objective of this study is to evaluate the effect of itraconazole on the pharmacokinetics of HS-20093 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, fixed-sequence, self-controlled clinical study designed to evaluate the effect of itraconazole on the pharmacokinetics of HS-20093 in patients with advanced solid tumors who have failed or are intolerant to standard therapy.

All participants will receive intravenous infusion of HS-20093 at a dose of 8 mg/kg every 3 weeks (Q3W), with each treatment cycle lasting 21 days. Participants will then take itraconazole capsules orally at 200 mg per dose during C2D17-C3D21

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced solid tumors that have failed standard therapy or are intolerant to standard treatment.
2. According to RECIST 1.1 criteria, participants must have at least one target lesion.
3. ECOG performance status score of 0-1 with no deterioration within 2 weeks prior to the first dose.
4. Minimum expected survival greater than 12 weeks.

Exclusion Criteria:

1. Patients with a contraindication for receiving itraconazole according to the prescribing information
2. Patients with severe, uncontrolled, or active cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Cmax of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Maximum concentration of HS-20093 and free toxin, measured by appropriate analytical methods.
AUC0-16d of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Area under the concentration-time curve from time zero to 16 days of HS-20093 and free free toxin, calculated by non-compartmental analysis.

SECONDARY OUTCOMES:
Tmax of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Time to reach maximum concentration of HS-20093 and free toxin, derived directly from observed concentration-time data.
t1/2 of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Terminal elimination half-life of HS-20093 and free toxin.
AUC0-∞ and AUC0-tau of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) and during the dosing interval (AUC0-tau) of HS-20093 and free toxin.
Cmin of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Minimum observed concentration of HS-20093 and free toxin.
CL of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Clearance of HS-20093 and free toxin.
V of HS-20093 and free toxin | Three treatment cycles, each cycle lasting for three weeks.
  Volume of distribution of HS-20093 and free toxin.
Incidence and severity of adverse events (AEs) | Screening to 90 days post-last dose
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a clinical study participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China